CLINICAL TRIAL: NCT06305312
Title: Community Services Navigation to Advance Health Equity in Breast Cancer Screening
Acronym: B-SINCERE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HCI166685; 1R01CA282409-01 (NIH)
Record Dates: First submitted 2024-02-29; First posted 2024-03-12 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): Standard referrals to community resources will be used for participants randomized to usual care.
  Interventions: Other: Usual Care
- Intervention (Experimental): Community Services Navigation with 211 Information Specialists (ISs) will conduct outreach to participants within 48 hours of referral through telephone, text, or email, depending on patient preference. Two weeks after initial contact ISs follow up with patients to provide additional support and document use of the referred services in ServicePoint.
  Interventions: Behavioral: Community Service Navigation

INTERVENTIONS:
Behavioral: Community Service Navigation — Patients randomized to the intervention will be directly referred to the United Way of Salt Lake's 211 community referral service for additional outreach.
  Arms: Intervention
Other: Usual Care — Standard referral to community resources.
  Arms: Usual Care

SUMMARY:
The goal of this study is to evaluate if adding community services navigation to the standard referral process for social needs is an effective and scalable strategy for addressing disparities in follow-up to abnormal breast cancer screening results. The investigators will determine the effectiveness of social needs referrals combined with a community services navigation intervention in the screening mammography setting to improving breast screening outcomes in underserved women.

DETAILED DESCRIPTION:
Disparities in breast cancer outcomes are persistent. In the United States, breast cancer is the most common, and second most deadly, cancer in women, with an estimated 281,550 new invasive breast cancer diagnoses and 43,600 breast cancer deaths in 2021. Underserved women, those who do not have adequate access to medical care, are represented disproportionately in those deaths, having lower incidence rates but higher mortality rates. While U.S. breast cancer mortality rates have decreased approximately 2% per year since 1990, socially and economically disadvantaged women have experienced increasing breast cancer mortality over that time. Rural women are more likely to experience diagnostic delays and are up to 1.5 times more likely to be diagnosed with advanced stages of disease compared with urban women.

Leveraging existing social systems for community navigation to facilitate breast screening follow-up. Our research has demonstrated that linkages between social needs screening in clinical settings and United Way 211's community referral service is possible using existing, low cost software solutions that can be adapted to clinical workflows. Specifically, the SINCERE 10-item social needs screener was combined with community services navigation and tested in a randomized controlled trial. That trial showed efficacy of the efficacy of this low cost, widely available solution to address the needs of vulnerable and underserved patients; namely, 211 active outreach v. passive information to address reported social needs. However, that trial was conducted in an Emergency Department, and has not been tested in other clinical settings. Building off of (collective) decades of work in breast cancer screening, the multiple PIs have formed an interdisciplinary team that has piloted an adaptation of the SINCERE social services screener (dubbed "B-SINCERE") in mammography clinics. This study will test the real-world efficacy (NIH stage 3) of the B-SINCERE community navigation intervention on increasing breast cancer screening episode completion. If efficacious, this intervention will be scalable with statewide community service providers and existing health information technology. Thus, the promise to make a real impact on early detection and improve breast cancer outcomes for underserved women with abnormal mammograms is the overarching driver of this work

ELIGIBILITY:
Inclusion Criteria:

* English and Spanish speakers
* Received an abnormal result of a screening mammogram
* Self-reports at least one social need on the B-SINCERE Screener

Exclusion Criteria:

* Patients who are currently in treatment for breast cancer
* Patients with a normal screening result.
* Patients who do not exhibit at least 1 social need according to their SINCERE screening result.
* Patients who don't speak English or Spanish
* Cognitive limitations that impede informed consent
* Patients living outside of Utah

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 1450 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Change in Social Needs | up to 18 months after baseline assessment
  Change in participants' level of social needs as measured by the B-SINCERE (Breast-Screener for Intensifying Community Referrals for Health) screener. To Test whether the use of a community services navigation intervention in conjunction with social service referrals decreases social needs compared to the referrals alone (usual care). B-SINCERE, reported on a 0-10 point scale, with 0=No Social Needs present, and 1-10=Social Needs present, anything greater than 0 indicates social needs and eligibility for the study.
Episode Completion (EC). | up to 18 months after baseline assessment
  EC is the name of a dichotomous scale, reported on a 2-point scale that is calculated from patient electronic health record (EHR), with 0=No Breast Cancer Screening completed, 1=Breast Cancer Screening completed.
  Impact of the community services navigation intervention on breast cancer screening episode completion and preventive care utilization among women with self-reported social needs. Preventive Care Utilization is a descriptive measure that is not reporting a score on a scale.

SECONDARY OUTCOMES:
Area deprivation index (ADI) | up to 18 months after baseline assessment
  DI is a tool for assessing an area's socioeconomic conditions. Scores range from 1-100, with lower scores indicating minimal socioeconomic disadvantage and higher scores indicating more socioeconomic disadvantage. This outcome measure will report ADI at 6 and 18 months of rural vs urban participants (based on ZIP codes) after baseline.
Rural Urban Commuting Area (RUCA) | up to 18 months after baseline assessment
  RUCA assesses urbanization, population density, and commuting. Scores range from 1 to 10, with lower scores indicating more urban areas and higher scores representing more rural areas. This outcome measure will report RUCA at 6 and 18 months of rural vs urban participants (based on ZIP codes) after baseline.
Social Service Utilization | up to 18 months after baseline assessment
  Social Service Utilization will assess how many study participants utilize 211 social services. This outcome measure will report the proportion of participants utilizing the following 211 medical care services: Finding healthy food, Adult education/job training/employment, Clothing/supplies, Housing, Transportation, Paying for health care, Paying bills, Child care, Other, 211 didn't help me get any services. This outcome measure will report social service utilization at 1, 6, and 18 months after the baseline assessment.
Breast cancer risk (Tyrer-Cuzick) | up to 18 months after baseline assessment
  The Tyrer-Cuzick breast cancer risk score estimates the likelihood of developing breast cancer. Scores range from 0 to 100 with lower scores indicating low breast cancer risk and high scores indicating high breast cancer risk. This outcome measure will report the mean breast cancer risk score at 6 and 18 months after the baseline assessment.
General Health Status | up to 18 months after baseline assessment
  General Health Status is a scale assessing general health. Scores range from 0 to 5, with lower scores indicating better health and higher scores indicating worse health. This outcome measure will report General Health Status at 1, 6, and 18 months after the baseline assessment.
Self-Report Generated Charlson Comorbidity Index | up to 18 months after baseline assessment
  Charlson Comorbidity Index is a score predicting mortality risk based on comorbidities. Scores range from 1 to 37, with lower scores indicating better mortality risk and higher scores representing worse mortality risk.
  This outcome measure will report the mean Charlson Comorbidity Index at 6 and 18 months after the baseline assessment.
Preventive services visits | from baseline assessment, up to 18 months
  Preventive services visits will measure how many participants complete their preventive visits. This outcome measure will report the proportion of participants who completed preventive visits such as the next annual mammogram, cervical cancer screening, or colorectal cancer screening. This outcome measure will report the proportion completing preventive services visits at 1, 6, and 18 months after the baseline assessment.
PROMIS Global Health | up to 18 months after baseline assessment
  PROMIS Global Health is a questionnaire assessing participants' health. Scores range from 0 to 32, with lower scores indicating worse health and higher scores indicating better health. This outcome measure will report PROMIS Global Health at 1, 6, and 18 months after the baseline assessment.
PROMIS Depression | up to 18 months after baseline assessment
  PROMIS Depression is a questionnaire assessing participants' mental health. Scores range from 0 to 32, with lower scores indicating better mental health and higher scores indicating worse mental health. This outcome measure will report PROMIS Depression at 1, 6, and 18 months after the baseline assessment.
Health Care Access | up to 18 months after baseline assessment
  Healthcare access is a 4-item questionnaire assessing patients' access to healthcare. Scores range from 0-12, with lower scores indicating worse access to healthcare and higher scores indicating better access to healthcare. This outcome measure will report Health Care Access at 6 and 18 months after the baseline assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Elissa Ozanne, PhD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- University of Utah Health Hospitals/Huntsman Cancer Institute Population Sciences, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cancer Stat Facts: Female Breast Cancer. 2022; https://seer.cancer.gov/statfacts/html/breast.html. Accessed Jul 11, 2022.
- [Background] Underserved group. Toolkit for Patient-Focused Therapy Development https://toolkit.ncats.nih.gov/glossary/underserved-group/. Accessed September 30, 2022.
- [Background] American Cancer Society. Cancer Facts & Figures for Hispanics/Latinos 2018-2020. Atlanta2018.
- [Background] Centers for Disease Control and Prevention National Center for Health Statistics. Death Rates for Selected Cancers by Race and Ethnicity, US, 2010-2014. 2016; https://www.cancer.org/content/dam/cancer-org/research/cancer-facts-and-statistics/annual-cancer-facts-and-figures/2017/death-rates-for-selected-cancers-by-race-and-ethnicity-us-2010-2014.pdf. Accessed Oct 11, 2021.
- [Background] Zahnd WE, James AS, Jenkins WD, Izadi SR, Fogleman AJ, Steward DE, Colditz GA, Brard L. Rural-Urban Differences in Cancer Incidence and Trends in the United States. Cancer Epidemiol Biomarkers Prev. 2018 Nov;27(11):1265-1274. doi: 10.1158/1055-9965.EPI-17-0430. Epub 2017 Jul 27. PMID 28751476
- [Background] Death Rates for Selected Cancers by Race and Ethnicity, US, 2010-2014. 2016; https://www.cancer.org/content/dam/cancer-org/research/cancer-facts-and-statistics/annual-cancer-facts-and-figures/2017/death-rates-for-selected-cancers-by-race-and-ethnicity-us-2010-2014.pdf. Accessed Oct 11, 2021.
- [Background] Henry KA, Sherman R, Farber S, Cockburn M, Goldberg DW, Stroup AM. The joint effects of census tract poverty and geographic access on late-stage breast cancer diagnosis in 10 US States. Health Place. 2013 May;21:110-21. doi: 10.1016/j.healthplace.2013.01.007. Epub 2013 Mar 1. PMID 23454732
- [Background] DeSantis CE, Ma J, Goding Sauer A, Newman LA, Jemal A. Breast cancer statistics, 2017, racial disparity in mortality by state. CA Cancer J Clin. 2017 Nov;67(6):439-448. doi: 10.3322/caac.21412. Epub 2017 Oct 3. PMID 28972651
- [Background] Doescher MP, Jackson JE. Trends in cervical and breast cancer screening practices among women in rural and urban areas of the United States. J Public Health Manag Pract. 2009 May-Jun;15(3):200-9. doi: 10.1097/PHH.0b013e3181a117da. PMID 19363399
- [Background] Roche LM, Niu X, Stroup AM, Henry KA. Disparities in Female Breast Cancer Stage at Diagnosis in New Jersey: A Spatial-Temporal Analysis. J Public Health Manag Pract. 2017 Sep/Oct;23(5):477-486. doi: 10.1097/PHH.0000000000000524. PMID 28430705
- [Background] Williams F, Jeanetta S, O'Brien DJ, Fresen JL. Rural-urban difference in female breast cancer diagnosis in Missouri. Rural Remote Health. 2015 Jul-Sep;15(3):3063. Epub 2015 Jul 29. PMID 26223824
- [Background] Vlahiotis A, Griffin B, Stavros AT, Margolis J. Analysis of utilization patterns and associated costs of the breast imaging and diagnostic procedures after screening mammography. Clinicoecon Outcomes Res. 2018 Mar 26;10:157-167. doi: 10.2147/CEOR.S150260. eCollection 2018. PMID 29618934
- [Background] Bleicher RJ. Timing and Delays in Breast Cancer Evaluation and Treatment. Ann Surg Oncol. 2018 Oct;25(10):2829-2838. doi: 10.1245/s10434-018-6615-2. Epub 2018 Jul 2. PMID 29968031
- [Background] Bleicher RJ, Ruth K, Sigurdson ER, Ross E, Wong YN, Patel SA, Boraas M, Topham NS, Egleston BL. Preoperative delays in the US Medicare population with breast cancer. J Clin Oncol. 2012 Dec 20;30(36):4485-92. doi: 10.1200/JCO.2012.41.7972. Epub 2012 Nov 19. PMID 23169513
- [Background] Bradley CJ, Given CW, Roberts C. Disparities in cancer diagnosis and survival. Cancer. 2001 Jan 1;91(1):178-88. doi: 10.1002/1097-0142(20010101)91:13.0.co;2-s. PMID 11148575
- [Background] Bradley CJ, Neumark D, Shickle LM, Farrell N. Differences in breast cancer diagnosis and treatment: experiences of insured and uninsured women in a safety-net setting. Inquiry. 2008 Fall;45(3):323-39. doi: 10.5034/inquiryjrnl_45.03.323. PMID 19069013
- [Background] Drake BF, Abadin SS, Lyons S, Chang SH, Steward LT, Kraenzle S, Goodman MS. Mammograms on-the-go-predictors of repeat visits to mobile mammography vans in St Louis, Missouri, USA: a case-control study. BMJ Open. 2015 Mar 20;5(3):e006960. doi: 10.1136/bmjopen-2014-006960. PMID 25795693
- [Background] Mizuguchi S, Barkley L, Rai S, Pan J, Roland L, Crawford S, Riley EC. Mobile Mammography, Race, and Insurance: Use Trends Over a Decade at a Comprehensive Urban Cancer Center. J Oncol Pract. 2015 Jan;11(1):e75-80. doi: 10.1200/JOP.2014.001477. Epub 2014 Nov 4. PMID 25371543
- [Background] Schunemann HJ, Lerda D, Quinn C, Follmann M, Alonso-Coello P, Rossi PG, Lebeau A, Nystrom L, Broeders M, Ioannidou-Mouzaka L, Duffy SW, Borisch B, Fitzpatrick P, Hofvind S, Castells X, Giordano L, Canelo-Aybar C, Warman S, Mansel R, Sardanelli F, Parmelli E, Grawingholt A, Saz-Parkinson Z, European Commission Initiative on Breast Cancer Contributor G. Breast Cancer Screening and Diagnosis: A Synopsis of the European Breast Guidelines. Ann Intern Med. 2019
- [Background] Bleicher RJ, Ruth K, Sigurdson ER, Beck JR, Ross E, Wong YN, Patel SA, Boraas M, Chang EI, Topham NS, Egleston BL. Time to Surgery and Breast Cancer Survival in the United States. JAMA Oncol. 2016 Mar;2(3):330-9. doi: 10.1001/jamaoncol.2015.4508. PMID 26659430
- [Background] Ashing-Giwa KT, Gonzalez P, Lim JW, Chung C, Paz B, Somlo G, Wakabayashi MT. Diagnostic and therapeutic delays among a multiethnic sample of breast and cervical cancer survivors. Cancer. 2010 Jul 1;116(13):3195-204. doi: 10.1002/cncr.25060. PMID 20564623
- [Background] Gorin SS, Heck JE, Cheng B, Smith SJ. Delays in breast cancer diagnosis and treatment by racial/ethnic group. Arch Intern Med. 2006 Nov 13;166(20):2244-52. doi: 10.1001/archinte.166.20.2244. PMID 17101943
- [Background] George P, Chandwani S, Gabel M, Ambrosone CB, Rhoads G, Bandera EV, Demissie K. Diagnosis and surgical delays in African American and white women with early-stage breast cancer. J Womens Health (Larchmt). 2015 Mar;24(3):209-17. doi: 10.1089/jwh.2014.4773. Epub 2015 Feb 4. PMID 25650628
- [Background] Elmore JG, Nakano CY, Linden HM, Reisch LM, Ayanian JZ, Larson EB. Racial inequities in the timing of breast cancer detection, diagnosis, and initiation of treatment. Med Care. 2005 Feb;43(2):141-8. doi: 10.1097/00005650-200502000-00007. PMID 15655427
- [Background] Ryu EB, Chang JM, Seo M, Kim SA, Lim JH, Moon WK. Tumour volume doubling time of molecular breast cancer subtypes assessed by serial breast ultrasound. Eur Radiol. 2014 Sep;24(9):2227-35. doi: 10.1007/s00330-014-3256-0. Epub 2014 Jun 4. PMID 24895040
- [Background] Neal RD, Tharmanathan P, France B, Din NU, Cotton S, Fallon-Ferguson J, Hamilton W, Hendry A, Hendry M, Lewis R, Macleod U, Mitchell ED, Pickett M, Rai T, Shaw K, Stuart N, Torring ML, Wilkinson C, Williams B, Williams N, Emery J. Is increased time to diagnosis and treatment in symptomatic cancer associated with poorer outcomes? Systematic review. Br J Cancer. 2015 Mar 31;112 Suppl 1(Suppl 1):S92-107. doi: 10.1038/bjc.2015.48. PMID 25734382
- [Background] Polverini AC, Nelson RA, Marcinkowski E, Jones VC, Lai L, Mortimer JE, Taylor L, Vito C, Yim J, Kruper L. Time to Treatment: Measuring Quality Breast Cancer Care. Ann Surg Oncol. 2016 Oct;23(10):3392-402. doi: 10.1245/s10434-016-5486-7. Epub 2016 Aug 8. PMID 27503492
- [Background] Kaufman CS, Shockney L, Rabinowitz B, Coleman C, Beard C, Landercasper J, Askew JB Jr, Wiggins D; Quality Initiative Committee. National Quality Measures for Breast Centers (NQMBC): a robust quality tool: breast center quality measures. Ann Surg Oncol. 2010 Feb;17(2):377-85. doi: 10.1245/s10434-009-0729-5. Epub 2009 Oct 16. PMID 19834768
- [Background] Comber H, Cronin DP, Deady S, Lorcain PO, Riordan P. Delays in treatment in the cancer services: impact on cancer stage and survival. Ir Med J. 2005 Sep;98(8):238-9. PMID 16255115
- [Background] Brazda A, Estroff J, Euhus D, Leitch AM, Huth J, Andrews V, Moldrem A, Rao R. Delays in time to treatment and survival impact in breast cancer. Ann Surg Oncol. 2010 Oct;17 Suppl 3:291-6. doi: 10.1245/s10434-010-1250-6. Epub 2010 Sep 19. PMID 20853049
- [Background] Ramachandran A, Snyder FR, Katz ML, Darnell JS, Dudley DJ, Patierno SR, Sanders MR, Valverde PA, Simon MA, Warren-Mears V, Battaglia TA; Patient Navigation Research Program Investigators. Barriers to health care contribute to delays in follow-up among women with abnormal cancer screening: Data from the Patient Navigation Research Program. Cancer. 2015 Nov 15;121(22):4016-24. doi: 10.1002/cncr.29607. Epub 2015 Aug 19. PMID 26385420
- [Background] Henderson LM, O'Meara ES, Haas JS, Lee CI, Kerlikowske K, Sprague BL, Alford-Teaster J, Onega T. The Role of Social Determinants of Health in Self-Reported Access to Health Care Among Women Undergoing Screening Mammography. J Womens Health (Larchmt). 2020 Nov;29(11):1437-1446. doi: 10.1089/jwh.2019.8267. Epub 2020 May 5. PMID 32366199
- [Background] Fallahian F, Nelson H, Pories S. The Role of Social Determinants of Health on Cancer Screening. 2022; https://www.facs.org/for-medical-professionals/news-publications/news-and-articles/bulletin/june-2022-volume-107-number-6/the-role-of-social-determinants-of-health-on-cancer-screening/.
- [Background] Alegria M, Araneta MR, Rivers B. The National Advisory Council on Minority Health and Health Disparities Reflection. Am J Public Health. 2019 Jan;109(S1):S14-S15. doi: 10.2105/AJPH.2019.304961. No abstract available. PMID 30699030
- [Background] Social Determinants of Health. Health topics 2022; https://www.who.int/health-topics/social-determinants-of-health#tab=tab_1. Accessed September 30, 2022.
- [Background] Centers for Disease Control and Prevention. Addressing Social Determinants of Health: Accelerating the Prevention and Control of HIV/AIDS, Viral Hepatitis, STD and TB. Atlanta, Georgia2009.
- [Background] Centers for Disease Control and Prevention. Centers for Disease Control and Prevention. Social Determinants of Health: Know What Affects Health. 2021; https://www.cdc.gov/socialdeterminants/.
- [Background] Maroko AR, Doan TM, Arno PS, Hubel M, Yi S, Viola D. Integrating Social Determinants of Health With Treatment and Prevention: A New Tool to Assess Local Area Deprivation. Prev Chronic Dis. 2016 Sep 15;13:E128. doi: 10.5888/pcd13.160221. PMID 27634778
- [Background] Phillips RL, Liaw W, Crampton P, Exeter DJ, Bazemore A, Vickery KD, Petterson S, Carrozza M. How Other Countries Use Deprivation Indices-And Why The United States Desperately Needs One. Health Aff (Millwood). 2016 Nov 1;35(11):1991-1998. doi: 10.1377/hlthaff.2016.0709. PMID 27834238
- [Background] DeMilto L, Nakashian M. Using social determinants of health data to improve health care and health: A learning report. Robert Wood Johnson Foundation. 2016;1:15
- [Background] Committee on Educating Health Professionals to Address the Social Determinants of Health; Board on Global Health; Institute of Medicine; National Academies of Sciences, Engineering, and Medicine. A Framework for Educating Health Professionals to Address the Social Determinants of Health. Washington (DC): National Academies Press (US); 2016 Oct 14. Available from http://www.ncbi.nlm.nih.gov/books/NBK395983/ PMID 27854400
- [Background] Garg A, Boynton-Jarrett R, Dworkin PH. Avoiding the Unintended Consequences of Screening for Social Determinants of Health. JAMA. 2016 Aug 23-30;316(8):813-4. doi: 10.1001/jama.2016.9282. No abstract available. PMID 27367226
- [Background] Henderson V, Tossas-Milligan K, Martinez E, Williams B, Torres P, Mannan N, Green L, Thompson B, Winn R, Watson KS. Implementation of an integrated framework for a breast cancer screening and navigation program for women from underresourced communities. Cancer. 2020 May 15;126 Suppl 10:2481-2493. doi: 10.1002/cncr.32843. PMID 32348565
- [Background] 211 Get Help Give Help. 2022; https://211utah.org/. Accessed September 30, 2022.
- [Background] Wallace AS, Luther B, Guo JW, Wang CY, Sisler S, Wong B. Implementing a Social Determinants Screening and Referral Infrastructure During Routine Emergency Department Visits, Utah, 2017-2018. Prev Chronic Dis. 2020 Jun 18;17:E45. doi: 10.5888/pcd17.190339. PMID 32553071
- [Background] Guo JW, Wallace AS, Luther BL, Wong B. Psychometric Evaluation of the Screener for Intensifying Community Referrals for Health. Eval Health Prof. 2022 Sep;45(3):270-276. doi: 10.1177/01632787211029360. Epub 2021 Jul 8. PMID 34235988
- [Background] Wallace AS, Luther BL, Sisler SM, Wong B, Guo JW. Integrating social determinants of health screening and referral during routine emergency department care: evaluation of reach and implementation challenges. Implement Sci Commun. 2021 Oct 7;2(1):114. doi: 10.1186/s43058-021-00212-y. PMID 34620248
- [Background] Sharareh N, Wallace AS, Brintz BJ, Wan N, Guo JW, Wong B. Associated factors with patient-reported unmet food needs among emergency department adult patients - A social need perspective. Prev Med Rep. 2022 Sep 7;29:101974. doi: 10.1016/j.pmedr.2022.101974. eCollection 2022 Oct. PMID 36161133
- [Background] MQSA National Statistics. 2022; https://www.fda.gov/radiation-emitting-products/mqsa-insights/mqsa-national-statistics. Accessed May 20, 2022.
- [Background] Aday LA, Andersen R. A framework for the study of access to medical care. Health Serv Res. 1974 Fall;9(3):208-20. PMID 4436074
- [Background] Andersen R, Bozzette S, Shapiro M, St Clair P, Morton S, Crystal S, Goldman D, Wenger N, Gifford A, Leibowitz A, Asch S, Berry S, Nakazono T, Heslin K, Cunningham W. Access of vulnerable groups to antiretroviral therapy among persons in care for HIV disease in the United States. HCSUS Consortium. HIV Cost and Services Utilization Study. Health Serv Res. 2000 Jun;35(2):389-416. PMID 10857469
- [Background] Andersen RM. Revisiting the behavioral model and access to medical care: does it matter? J Health Soc Behav. 1995 Mar;36(1):1-10. PMID 7738325
- [Background] Andersen RM, Davidson PL. Improving access to care in America. Changing the US Health Care System. 2nd ed. San Fransisco: Josey-Bass; 2001.
- [Background] Gelberg L, Andersen RM, Leake BD. The Behavioral Model for Vulnerable Populations: application to medical care use and outcomes for homeless people. Health Serv Res. 2000 Feb;34(6):1273-302. PMID 10654830
- [Background] Phillips KA, Morrison KR, Andersen R, Aday LA. Understanding the context of healthcare utilization: assessing environmental and provider-related variables in the behavioral model of utilization. Health Serv Res. 1998 Aug;33(3 Pt 1):571-96. PMID 9685123
- [Background] Miller KA, Hillier D, Russ C, Luercio M, Winn AS. Applying Self-Determination Theory to Redesign an Inpatient Care Team. Acad Pediatr. 2019 Apr;19(3):351-353. doi: 10.1016/j.acap.2018.09.010. Epub 2018 Oct 9. No abstract available. PMID 30312681
- [Background] Partelow S. A review of the social-ecological systems framework: applications, methods, modifications, and challenges. Ecology and Society. 2018;23(4)
- [Background] Henderson LM, Hubbard RA, Zhu W, Weiss J, Wernli KJ, Goodrich ME, Kerlikowske K, DeMartini W, Ozanne EM, Onega T. Preoperative Breast Magnetic Resonance Imaging Use by Breast Density and Family History of Breast Cancer. J Womens Health (Larchmt). 2018 Aug;27(8):987-993. doi: 10.1089/jwh.2017.6428. Epub 2018 Jan 15. PMID 29334616
- [Background] Onega T, Weiss JE, Goodrich ME, Zhu W, DeMartini WB, Kerlikowske K, Ozanne E, Tosteson ANA, Henderson LM, Buist DSM, Wernli KJ, Herschorn SD, Hotaling E, O'Donoghue C, Hubbard R. Relationship between preoperative breast MRI and surgical treatment of non-metastatic breast cancer. J Surg Oncol. 2017 Dec;116(8):1008-1015. doi: 10.1002/jso.24796. Epub 2017 Nov 11. PMID 29127715
- [Background] Ozanne EM, Weiss JE, Onega T, DeMartini W, Kerlikowske K, Buist DS, Henderson L, Hubbard RA, Goodrich M, Tosteson AN, Virnig BA, O'Donoghue C. Locoregional treatment of breast cancer in women with and without preoperative magnetic resonance imaging. Am J Surg. 2017 Jan;213(1):132-139.e2. doi: 10.1016/j.amjsurg.2016.03.014. Epub 2016 Jun 12. PMID 27421187
- [Background] Ballard-Barbash R, Taplin SH, Yankaskas BC, Ernster VL, Rosenberg RD, Carney PA, Barlow WE, Geller BM, Kerlikowske K, Edwards BK, Lynch CF, Urban N, Chrvala CA, Key CR, Poplack SP, Worden JK, Kessler LG. Breast Cancer Surveillance Consortium: a national mammography screening and outcomes database. AJR Am J Roentgenol. 1997 Oct;169(4):1001-8. doi: 10.2214/ajr.169.4.9308451. No abstract available.
- [Background] Incidence Rate Report for Utah by County, Breast (Late Stage), 2014-2018, White Non-Hispanic, Female, All Ages. https://statecancerprofiles.cancer.gov/incidencerates/index.php?stateFIPS=49&areatype=county&cancer=055&race=07&sex=2&age=001&stage=211&year=0&type=incd&sortVariableName=rate&sortOrder=default&output=0#results. Accessed Oct 11, 2021.
- [Background] Onega T, Tosteson TD, Weiss J, Haas JS, Goodrich M, DiFlorio R, Brackett C, Clark C, Harris K, Tosteson ANA. Multi-level Influences on Breast Cancer Screening in Primary Care. J Gen Intern Med. 2018 Oct;33(10):1729-1737. doi: 10.1007/s11606-018-4560-1. Epub 2018 Aug 3. PMID 30076569
- [Background] Beaber EF, Sprague BL, Tosteson ANA, Haas JS, Onega T, Schapira MM, McCarthy AM, Li CI, Herschorn SD, Lehman CD, Wernli KJ, Barlow WE. Multilevel Predictors of Continued Adherence to Breast Cancer Screening Among Women Ages 50-74 Years in a Screening Population. J Womens Health (Larchmt). 2019 Aug;28(8):1051-1059. doi: 10.1089/jwh.2018.6997. Epub 2018 Nov 27. PMID 30481098
- [Background] Schapira MM, Barlow WE, Conant EF, Sprague BL, Tosteson ANA, Haas JS, Onega T, Beaber EF, Goodrich M, McCarthy AM, Herschorn SD, Skinner CS, Harrington TO, Geller B. Communication Practices of Mammography Facilities and Timely Follow-up of a Screening Mammogram with a BI-RADS 0 Assessment. Acad Radiol. 2018 Sep;25(9):1118-1127. doi: 10.1016/j.acra.2017.12.028. Epub 2018 Feb 9. PMID 29433892
- [Background] Buist DSM, Gao H, Anderson ML, Onega T, Brandzel S, Rabelhofer MA, Bradford SC, Aiello Bowles EJ. Breast cancer screening outreach effectiveness: Mammogram-specific reminders vs. comprehensive preventive services birthday letters. Prev Med. 2017 Sep;102:49-58. doi: 10.1016/j.ypmed.2017.06.028. Epub 2017 Jun 24. PMID 28655547
- [Background] Lee CI, Zhu W, Onega T, Henderson LM, Kerlikowske K, Sprague BL, Rauscher GH, O'Meara ES, Tosteson ANA, Haas JS, diFlorio-Alexander R, Kaplan C, Miglioretti DL. Comparative Access to and Use of Digital Breast Tomosynthesis Screening by Women's Race/Ethnicity and Socioeconomic Status. JAMA Netw Open. 2021 Feb 1;4(2):e2037546. doi: 10.1001/jamanetworkopen.2020.37546. PMID 33606032
- [Background] Ozanne EM, Klemp JR, Esserman LJ. Breast cancer risk assessment and prevention: a framework for shared decision-making consultations. Breast J. 2006 Mar-Apr;12(2):103-13. doi: 10.1111/j.1075-122X.2006.00217.x. PMID 16509834
- [Background] Euhus DM. Breast cancer prevention in the 21st century: defining the challenge. Breast J. 2006 Mar-Apr;12(2):97-8. doi: 10.1111/j.1075-122X.2006.00215.x. No abstract available. PMID 16509832
- [Background] Ozanne EM, Annis C, Adduci K, Showstack J, Esserman L. Pilot trial of a computerized decision aid for breast cancer prevention. Breast J. 2007 Mar-Apr;13(2):147-54. doi: 10.1111/j.1524-4741.2007.00395.x. PMID 17319855
- [Background] Ozanne EM, Howe R, Omer Z, Esserman LJ. Development of a personalized decision aid for breast cancer risk reduction and management. BMC Med Inform Decis Mak. 2014 Jan 14;14:4. doi: 10.1186/1472-6947-14-4. PMID 24422989
- [Background] Ozanne EM, Schneider KH, Soeteman D, Stout N, Schrag D, Fordis M, Punglia RS. onlineDeCISion.org: a web-based decision aid for DCIS treatment. Breast Cancer Res Treat. 2015 Nov;154(1):181-90. doi: 10.1007/s10549-015-3605-y. PMID 26475704
- [Background] Ozanne EM, Soeteman DI, Frank ES, Clarke J, Hassett MJ, Stout NK, Punglia RS. Commentary: Creating a patient-centered decision aid for ductal carcinoma in situ. Breast J. 2020 Jul;26(7):1498-1499. doi: 10.1111/tbj.13779. Epub 2020 Feb 8. No abstract available. PMID 32034829
- [Background] Cancer Screening and Education Bus. Cancer Screening & Prevention https://healthcare.utah.edu/huntsmancancerinstitute/screening-prevention/mobile-screening.php. Accessed September 30, 2022.
- [Background] Chew LD, Bradley KA, Boyko EJ. Brief questions to identify patients with inadequate health literacy. Fam Med. 2004 Sep;36(8):588-94. PMID 15343421
- [Background] Chew LD, Griffin JM, Partin MR, Noorbaloochi S, Grill JP, Snyder A, Bradley KA, Nugent SM, Baines AD, Vanryn M. Validation of screening questions for limited health literacy in a large VA outpatient population. J Gen Intern Med. 2008 May;23(5):561-6. doi: 10.1007/s11606-008-0520-5. Epub 2008 Mar 12. PMID 18335281
- [Background] Sarkar U, Schillinger D, Lopez A, Sudore R. Validation of self-reported health literacy questions among diverse English and Spanish-speaking populations. J Gen Intern Med. 2011 Mar;26(3):265-71. doi: 10.1007/s11606-010-1552-1. Epub 2010 Nov 6. PMID 21057882
- [Background] Warwick J, Birke H, Stone J, Warren RM, Pinney E, Brentnall AR, Duffy SW, Howell A, Cuzick J. Mammographic breast density refines Tyrer-Cuzick estimates of breast cancer risk in high-risk women: findings from the placebo arm of the International Breast Cancer Intervention Study I. Breast Cancer Res. 2014 Oct 8;16(5):451. doi: 10.1186/s13058-014-0451-5. PMID 25292294
- [Background] Charlson M, Szatrowski TP, Peterson J, Gold J. Validation of a combined comorbidity index. J Clin Epidemiol. 1994 Nov;47(11):1245-51. doi: 10.1016/0895-4356(94)90129-5. PMID 7722560
- [Background] Hailu D, Asnake. Guidelines for Using Rural-Urban Classification Systems for Community Health Assessment. In: Health WSDo, ed: Washington State Department of Health; 2016:1-26.
- [Background] Knighton AJ, Savitz L, Belnap T, Stephenson B, VanDerslice J. Introduction of an Area Deprivation Index Measuring Patient Socioeconomic Status in an Integrated Health System: Implications for Population Health. EGEMS (Wash DC). 2016 Aug 11;4(3):1238. doi: 10.13063/2327-9214.1238. eCollection 2016. PMID 27683670
- [Background] Onega T, Haas JS, Bitton A, Brackett C, Weiss J, Goodrich M, Harris K, Pyle S, Tosteson AN. Alignment of breast cancer screening guidelines, accountability metrics, and practice patterns. Am J Manag Care. 2017 Jan;23(1):35-40. PMID 28141929
- [Background] Schiffelbein JE, Carluzzo KL, Hasson RM, Alford-Teaster JA, Imset I, Onega T. Barriers, Facilitators, and Suggested Interventions for Lung Cancer Screening Among a Rural Screening-Eligible Population. J Prim Care Community Health. 2020 Jan-Dec;11:2150132720930544. doi: 10.1177/2150132720930544. PMID 32506999
- [Background] Raffin E, Onega T, Bynum J, Austin A, Carmichael D, Bronner K, Goodney P, Hyams ES. Are there regional tendencies toward controversial screening practices? A study of prostate and breast cancer screening in a Medicare population. Cancer Epidemiol. 2017 Oct;50(Pt A):68-75. doi: 10.1016/j.canep.2017.07.015. Epub 2017 Aug 17. PMID 28822325
- [Background] Haas J, Schapira M, Sprague B, Tosteson A, Klabunde C, Chen J, Bitton A, Beaber E, Onega T, Kim J, MacLean C. Changes in Primary Care Practice Following New USPSTF Breast and Cervical Cancer Screening Guidelines. AcademyHealth 2015 Annual Research Meeting; June 15, 2015.
- [Background] National Cancer Institute Division of Cancer Control & Population Sciences. Population-based Research to Optimize the Screening Process (PROSPR). 2021; https://healthcaredelivery.cancer.gov/prospr/prospr1/.
- [Background] Cozzi A, Schiaffino S, Giorgi Rossi P, Sardanelli F. Breast cancer screening: in the era of personalized medicine, age is just a number. Quant Imaging Med Surg. 2020 Dec;10(12):2401-2407. doi: 10.21037/qims-2020-26. No abstract available. PMID 33269240
- [Background] Tosteson AN, Beaber EF, Tiro J, Kim J, McCarthy AM, Quinn VP, Doria-Rose VP, Wheeler CM, Barlow WE, Bronson M, Garcia M, Corley DA, Haas JS, Halm EA, Kamineni A, Rutter CM, Tosteson TD, Trentham-Dietz A, Weaver DL; PROSPR consortium. Variation in Screening Abnormality Rates and Follow-Up of Breast, Cervical and Colorectal Cancer Screening within the PROSPR Consortium. J Gen Intern Med. 2016 Apr;31(4):372-9. doi: 10.1007/s11606-015-3552-7. PMID 26658934
- [Background] Baum JK, Hanna LG, Acharyya S, Mahoney MC, Conant EF, Bassett LW, Pisano ED. Use of BI-RADS 3-probably benign category in the American College of Radiology Imaging Network Digital Mammographic Imaging Screening Trial. Radiology. 2011 Jul;260(1):61-7. doi: 10.1148/radiol.11101285. Epub 2011 Apr 18. PMID 21502382
- [Background] Breast Imaging Reporting & Data System (BI-RADS (R)). 2013; https://www.acr.org/Clinical-Resources/Reporting-and-Data-Systems/Bi-Rads. Accessed July 25, 2022.
- [Background] Bevers TB, Anderson BO, Bonaccio E, Buys S, Daly MB, Dempsey PJ, Farrar WB, Fleming I, Garber JE, Harris RE, Heerdt AS, Helvie M, Huff JG, Khakpour N, Khan SA, Krontiras H, Lyman G, Rafferty E, Shaw S, Smith ML, Tsangaris TN, Williams C, Yankeelov T; National Comprehensive Cancer Network. NCCN clinical practice guidelines in oncology: breast cancer screening and diagnosis. J Natl Compr Canc Netw. 2009 Nov;7(10):1060-96. doi: 10.6004/jnccn.2009.0070. No abstract available. PMID 19930975
- [Background] Guest G, MacQueen KM, Namey EE. Applied Thematic Analysis. SAGE Publications, Inc.; 2012.
- [Background] Glaser BG, Strauss AL. Discovery of Grounded Theory: Strategies for Qualitative Research. Routledge; 2017.
- [Background] Krippendorff K. Quantitative guidelines for communicable disease control programs. Biometrics. 1978 Mar;34(1):142. No abstract available. PMID 630036
- [Background] Morse JM. The Significance of Saturation. Qualitative Health Research. 1995;5(2):147-149
- [Background] Guest G, Bunce A, Johnson L. How Many Interviews Are Enough?:An Experiment with Data Saturation and Variability. Field Methods. 2006;18(1):59-82
- [Background] Center for HOPE. 2022; https://healthcare.utah.edu/huntsmancancerinstitute/about-us/center-for-hope.php. Accessed September 30, 2022.
- [Background] Center for HOPE. Huntsman Cancer Institute Research 2022; https://uofuhealth.utah.edu/huntsman/labs/center-for-hope. Accessed September 30, 2022.
- [Derived] Beck K, Mitchell M, Wallace AS, Freer PE, Wong B, Kepka D, Watt MH, McNall S, Kolomaya A, Ariotti A, Mulford M, Onega T, Ozanne EM. Community navigation intervention for social needs in patients with abnormal mammography: a randomized controlled trial study protocol. BMC Public Health. 2025 Aug 26;25(1):2926. doi: 10.1186/s12889-025-24372-x. PMID 40859259